CLINICAL TRIAL: NCT07214363
Title: Malignant Liver Tumors Who Are Unsuitable for Surgical Resection, Irreversible Electroporation (IRE) Ablation Will be Performed for Tumors Located Adjacent to Blood Vessels.
Brief Title: The Safety and Efficacy of Irreversible Electroporation for the Treatment of Perivascular Liver Cancers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202309001DIPC
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Liver Cancer; Ablation Techniques; Radiology
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- liver tumors are unsuitable for surgical resection (Experimental): Participants with liver cancer, considered for local treatment of liver tumors of size measuring <5 cm and without any signs of extra-hepatic metastasis, will be enrolled to be treated
  Interventions: Device: Irreversible Electroporation Ablation Generator

INTERVENTIONS:
Device: Irreversible Electroporation Ablation Generator — The irreversible electroporation ablation system (Irreversible Electroporation Ablation Generator) used in this study delivers an ablation field with a voltage of 3,000 volts. It received U.S. Food and Drug Administration (FDA) approval in 2023 but has not yet been introduced in Taiwan. This study will target participants with malignant liver tumors who are unsuitable for surgical resection but are eligible for local ablation therapy, specifically those with tumors located adjacent to the inferior vena cava, hepatic veins, or within 1 cm of the main trunks of both portal veins. A total of 20 participants will undergo ablation treatment under intubation and general anesthesia. Postoperative monitoring will focus on potential complications, and participants will be followed for four months to assess complete tumor ablation and intrahepatic recurrence, in order to verify the clinical feasibility and advantages of this system.

SUMMARY:
Malignant liver tumors are among the most common cancers worldwide, with over 10,000 new cases reported annually in Taiwan. Despite the availability of various treatment options, the prognosis for primary hepatocellular carcinoma and other metastatic liver cancers remains poor, with more than 8,000 deaths each year. The majority of patients (approximately 70%-85%) are diagnosed at an advanced stage or are deemed unresectable. In contrast, patients with small tumors often have a chance of cure. According to numerous studies, patients undergoing hepatic resection achieve a five-year disease-free survival rate exceeding 50%.

For patients with unresectable malignant liver tumors who do not have vascular invasion or extrahepatic metastasis, radiofrequency ablation (RFA) serves as an alternative curative treatment. However, a major limitation of RFA lies in its reduced efficacy when tumors are located near blood vessels, making complete ablation difficult. Irreversible electroporation (IRE) offers a safer ablation modality that is unaffected by vascular proximity. Both preclinical and clinical studies have demonstrated that IRE is a safe and effective treatment for liver tumors. According to reports in the international journal Radiology, complete ablation rates of 77.3%-92% have been achieved in patients with liver cancer treated with IRE, with complication rates of around 19%, most of which were mild.

The irreversible electroporation ablation system (Irreversible Electroporation Ablation Generator) used in this study delivers an ablation field with a voltage of 3,000 volts. It received U.S. Food and Drug Administration (FDA) approval in 2023 but has not yet been introduced in Taiwan. This study will target patients with malignant liver tumors who are unsuitable for surgical resection but are eligible for local ablation therapy, specifically those with tumors located adjacent to the inferior vena cava, hepatic veins, or within 1 cm of the main trunks of both portal veins. A total of 20 patients will undergo ablation treatment under intubation and general anesthesia. Postoperative monitoring will focus on potential complications, and patients will be followed for four months to assess complete tumor ablation and intrahepatic recurrence, in order to verify the clinical feasibility and advantages of this system.

ELIGIBILITY:
Inclusion Criteria:

* Malignant liver cancer including hepatocellular carcinoma (HCC), cholangiocarcinoma and metastatic liver cancers, The diagnosis of cholangiocarcinoma or metastatic liver cancers with pathologic proven, and the diagnosis of HCC will be made by pathology / cytology or according to the AASLD (2018) diagnostic criteria. In brief, Nodules larger than 1 cm found on ultrasound screening of a cirrhotic liver should be investigated further with either tri-phase multidetector CT scan or dynamic contrast enhanced MRI. If the appearances are typical of HCC (i.e., hypervascular in the arterial phase with washout in the portal venous or delayed phase), the lesion should be treated as HCC. If the findings are not characteristic or the vascular profile is not typical, a second contrast enhanced study with the other imaging modality should be performed, or the lesion should be biopsied. Biopsies of small lesions should be evaluated by expert pathologists. Tissue that is not clearly HCC should be stained with all the available markers including CD34, CK7, glypican 3, HSP-70, and glutamine synthetase to improve diagnostic accuracy.
* Unsuitable for surgical resection but local ablation is indicated, however, the distance between tumour and inferior vena cava, hepatic veins or bilateral; portal veins is smaller than 1 cm.
* The patient can tolerate endotracheal intubation and general anaesthesia.
* The tumour number is less than or equal to 3,
* Maximal tumor size must be ≤ 5 cm in diameter,
* Child-Pugh class A-B,
* Eastern Cooperative Oncology Group (ECOG) score of 0-1,
* American Society of Anesthesiologists (ASA) score ≤ 3,
* Adequate bone marrow and liver function (1). PT-INR ≦ 2.0. (2). Platelet count ≥ 100 K/Μl (3). Total bilirubin ≦ 3 mg/dL (4). ALT and AST < 5 x upper limit of normal
* Prior Informed Consent Form
* Life expectancy of at least 3 months.

Exclusion Criteria:

-History of cardiac disease: (A)Congestive heart failure >NYHA class 2; (B)Active Coronary Artery Disease (defined as myocardial infarction within 6 months prior to screening); (C)Cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker (beta blockers are permitted)

* Immunotherapy or chemotherapy ≤ 6 weeks prior to the procedure;
* Contraindicated to abdominal CT and MRI
* Allergy to muscle relaxant.
* History of epilepsy
* Women who are pregnant or women of child-bearing potential without using an acceptable method of contraception,
* Patients received treatment with an investigational agent/ procedure within 30 days.
* Patients with hypertension or arrythmia under poor medical control
* Acute infection or inflammation, acute and severe dysfunction of heart, liver and kidney, and the patients with metallic implantation including pacemaker.
* Known history of HIV infection
* Concurrent extrahepatic cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the efficacy of irreversible electroporation for the treatment of primary or secondary liver cancers in participants who are not suitable candidates for surgical intervention. | 1 month
  The primary measure for this will be the evaluation of tumor response according to the modified RECIST criteria by CT or MR imaging performed

SECONDARY OUTCOMES:
Safety using the CTCAE Version 4.0 criteria | 4 months
local tumor recurrences | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan